CLINICAL TRIAL: NCT02580409
Title: Maintaining Physical Independence in Older Adults
Brief Title: REACH Pilot Study (Rehabilitation Enhancing Aging Through Connected Health)
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Boston University (Other); Brandeis University (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jonathan F. Bean, MD, MS, MPH, MD, MS, MPH, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000393
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Mobility Limitation
Keywords: health care utilization; health care costs
MeSH Terms: conditions — Mobility Limitation; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm studies (Other): Behavioral Intervention
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Investigators are proposing an innovative rehabilitative care program for older primary care patients at risk for mobility decline. The program targets newly identified risk factors for mobility decline and utilizes mobile health technology to deliver patient centered care more efficiently. Study participants will receive exercise instruction with a licensed physical therapist for an average of 8-10 training sessions, with the possibility of up to 16 sessions. some at home and some in the clinic. The exercise training sessions will focus on improving mobility, balance and ability to get up from a chair with the use of an exercise application (Wellpepper) being used on a study issued iPad.

SUMMARY:
Rehabilitation Enhancing Aging through Connected Health, REACH, is designed to evaluate the benefits of a novel rehabilitative care program on physical function utilizing mobile health technology to deliver patient centered care more efficiently and health care utilization after one year of follow up.

DETAILED DESCRIPTION:
Rehabilitation Enhancing Aging through Connected Health, REACH, is designed to evaluate the benefits of a novel rehabilitative care program on physical function utilizing mobile health technology to deliver patient centered care more efficiently and health care utilization after one year of follow up. Study staff will recruit 76 community dwelling older adult primary care patients. The same procedures that were approved by the IRB for the Boston RISE cohort study. This study was initiated in 2009 and its data is publicly archived. will be used for REACH recruitment, screening and enrollment of potential participants. This process will be centered at Spaulding Cambridge Outpatient Clinic (SCOC). Potential participants will be contacted and a brief phone screen will be conducted. Eligible and interested participants will be scheduled for the consent/screen visit. If the participant consents, the study staff will administer three tests to determine final eligibility for study involvement. These include: Mini Mental Status Exam, the Short Physical Performance Battery (SPPB) and the Long Distance Corridor Walk.

Qualified participants will complete all baseline and 1-year assessments at SCOC. The assessments include: the Late Life Function and Disability Index (LLFDI), Hopkins Verbal Learning Test, Trail Making, Digit Symbol Substitution Test, Katz Comorbidity, depression (PHQ-9), Activities Specific Balance Scale, Barriers Specific Self-Efficacy Scale, Computer Attitude Scale, McGill Pain Map, Brief Pain Inventory, Figure 8 walk test, grip strength testing, single leg press strength and speed testing, ankle/knee ROM, the trunk extensor endurance test and stair climb power test.

The exercise/technology training with a licensed physical therapist will consist of 8-10 (with the possibility of up to 16 sessions) clinic or home visits interspersed over a 9-month period and will take place after baseline at one of two locations per choice of participant: SCOC or BU Center for Neurorehabilitation. During the clinic/home visits, the assigned exercises are video recorded using the Wellpepper clinician version housed on an iPad mini. During and after the in-person visits, the PTs will remotely monitor exercise adherence, provide feedback, progress the exercise program and answer participants' questions using the chat feature of the exercise app. PT support will be tapered over the course of this 9-month period as the participants become more successful at integrating exercise into their lives using the provided technology. Over the final 3 months of the study, participants will continue to perform exercises independently with reduced PT involvement. PT support will be available through the chat feature if participants have questions or concerns.

Participants will be contacted at quarterly intervals and asked to self-report recent falls, hospitalizations, ER visits and PT (outside of their participation in this study). At 6 months the LLFDI will be administered over the phone. In addition, the PT will perform these performance based assessments during a clinic visit: SPPB, ankle/knee ROM, trunk extensor endurance test and the stair climb power test.

Collaborators at Brandeis University will access CMS claims data for all participants during the year of participation and for an additional six months after study participation ends to evaluate health care utilization and health care costs after 1-year of follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 65-95 years
2. Able to understand and communicate in English
3. Difficulty or task modification with walking ½ mile (6 blocks) or climbing one flight of stairs
4. Ability to continuously walk 400 m in less than 15 minutes without stopping for more than a minute at a time, sitting, leaning, or the help of another person
5. Lives in a zip code within 10 mile radius of Spaulding Cambridge Facility
6. Baseline Short Physical Performance Battery (SPPB) scores from 3-12 with <20% of SPPB scores in the 11-12 range

Exclusion Criteria:

1. Presence of a terminal disease (e.g. receiving hospice services, metastatic cancer)
2. Major surgery or Myocardial Infarction in the last 6 months
3. Planned major surgery (e.g. joint replacement)
4. Planned move from the Boston area within 1.5 years
5. Mini-mental state exam (MMSE) score <20
6. Major medical problems interfering with safe and successful testing (examples may include: history hip replacement with recurrent dislocation, uncontrolled hypertension, use of supplemental oxygen)

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan F Bean, MD, MS, MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital Cambridge, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Bean JF, Brown L, DeAngelis TR, Ellis T, Kumar VSS, Latham NK, Lawler D, Ni M, Perloff J. The Rehabilitation Enhancing Aging Through Connected Health Prehabilitation Trial. Arch Phys Med Rehabil. 2019 Nov;100(11):1999-2005. doi: 10.1016/j.apmr.2019.04.015. Epub 2019 May 29. PMID 31152705
- [Derived] Ni M, Brown LG, Lawler D, Ellis TD, Deangelis T, Latham NK, Perloff J, Atlas SJ, Percac-Lima S, Bean JF. The rehabilitation enhancing aging through connected health (REACH) study: study protocol for a quasi-experimental clinical trial. BMC Geriatr. 2017 Sep 20;17(1):221. doi: 10.1186/s12877-017-0618-x. PMID 28931377

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single-arm Studies
Started | 75
Completed | 68
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Single-arm Studies
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.4 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 55
  More than one race | 0
  Unknown or Not Reported | 4
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 27.5 (4.39)

OUTCOME MEASURES:

1. Primary Outcome: Change in Late Life Function and Disability Index (Function Domain Only)
Description: The Late-Life Function & Disability Instrument (Late-Life FDI) is a self-report evaluative outcome instrument for community-dwelling older adults. It is designed to assess and be responsive to meaningful change in two distinct outcomes: function and disability. It is possible to measure one without the other. For this study, only the functional domain will be used. Functional limitations pertain to limitations in a person's ability to do discrete actions or activities. This domain is scaled between 0-100 with higher scores reflecting better mobility.
  The outcome measure is presented as a coefficient of change within a regression model evaluating baseline and follow up values of the outcome..
Time Frame: Assessed at baseline visit and 12 months after baseline visit (1 year visit)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single-arm Studies
Number analyzed (Participants) | 68
units on a scale | 1.67 (.55)

2. Other Pre Specified Outcome: Change in the Short Physical Performance Battery (SPPB)
Description: The Short Physical Performance Battery (SPPB) is an objective physical performance assessment tool for evaluating lower extremity functioning in older persons.
Time Frame: Assessed at screen visit, 6 month assessment after baseline visit and 12 months after baseline visit (1 year visit)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Single-arm Studies
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT02580409/Prot_SAP_000.pdf